CLINICAL TRIAL: NCT05552976
Title: A Phase 3, Two-stage, Randomized, Multicenter, Open-label Study Comparing Mezigdomide (CC-92480/BMS-986348), Carfilzomib, and Dexamethasone (MeziKD) Versus Carfilzomib and Dexamethasone (Kd) in Participants With Relapsed or Refractory Multiple Myeloma (RRMM): SUCCESSOR-2
Brief Title: A Study to Evaluate Mezigdomide in Combination With Carfilzomib and Dexamethasone (MeziKD) Versus Carfilzomib and Dexamethasone (Kd) in Participants With Relapsed or Refractory Multiple Myeloma (SUCCESSOR-2)
Acronym: SUCCESSOR-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA057-008
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: BMS-986348; CC-92480; Carfilzomib; Dexamethasone; Multiple Myeloma; Mezigdomide
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: This is a two-stage inferentially seamless design.
Masking Description: This is an open-label study; however, any review of aggregate study data by the Sponsor will be performed in a blinded manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MeziKd (Mezigdomide + Carfilzomib + Dexamethasone) (Experimental)
  Interventions: Drug: Mezigdomide; Drug: Carfilzomib; Drug: Dexamethasone
- Kd (Carfilzomib + Dexamethasone) (Active Comparator)
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480
  Arms: MeziKd (Mezigdomide + Carfilzomib + Dexamethasone)
Drug: Carfilzomib — Specified dose on specified days
  Other Names: Kyprolis
Drug: Dexamethasone — Specified dose on specified days
  Other Names: Decadron; Dex

SUMMARY:
The purpose of the study is to compare Mezigdomide (CC-92480/BMS-986348) with carfilzomib and dexamethasone (MeziKD) against carfilzomib and dexamethasone (Kd) in the treatment of RRMM: SUCCESSOR-2.

ELIGIBILITY:
Inclusion Criteria

- Participant has documented diagnosis of multiple myeloma and measurable disease, defined as any of the following:.

i) Myeloma-protein (M-protein) ≥ 0.5 grams/deciliter (g/dL) by serum protein electrophoresis (sPEP), or.

ii) M-protein ≥ 200 milligrams (mg)/24-hour urine collection by urine protein electrophoresis (uPEP) or,.

iii) For participants without measurable disease in sPEP or uPEP: serum free light chain levels > 100 mg/liter (L) (10 mg/dL) involved light chain and an abnormal κ/λ free light chain ratio.

* Participant has received at least one prior line of anti-myeloma therapy. Note: One line can contain several phases (e.g., induction, [with or without] hematopoietic stem cell transplant, (with or without) consolidation, and/or [with or without] maintenance therapy).
* Participant must have received prior treatment with lenalidomide and at least 2 cycles of an anti-CD38 monoclonal antibody (mAb) (participants who were intolerant of an anti-CD38 mAb and received < 2 cycles are still eligible).
* Participant achieved minimal response or better to at least 1 prior anti-myeloma therapy.
* Participant must have documented disease progression during or after their last antimyeloma regimen.

Exclusion Criteria

* Participant who has had prior treatment with mezigdomide or carfilzomib.
* Participant has previously received allogeneic stem cell transplant at any time or received autologous stem cell transplant within 12 weeks of initiating study treatment.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2029-07-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 5 years

SECONDARY OUTCOMES:
Recommended Mezigdomide Dose | Up to 12 months
  Stage 1 only
Plasma concentrations of Mezigdomide in Combination with Carfilzomib and Dexamethasone | Up to 176 days
  Stage 1 only
Overall Survival (OS) | Up to approximately 5 years
Overall Response (OR) | Up to approximately 5 years
Rate Of Very Good Partial Response (VGPR) Or Better (VGPRR) | Up to approximately 5 years
  VGPRR will be calculated as the percentage of participants who achieve best response of VGPR or better according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma.
Complete Response (CR) Or Better (CRR) | Up to approximately 5 years
  CRR will be calculated as the percentage of participants who achieve best response of CR or better according to the IMWG Uniform Response Criteria for Multiple Myeloma.
Time To Response (TTR) | Up to approximately 5 years
Duration Of Response (DOR) | Up to approximately 5 years
Time To Progression (TTP) | Up to approximately 5 years
Time To Next Treatment (TTNT) | Up to approximately 5 years
Progression-free Survival 2 (PFS-2) | Up to approximately 5 years
Minimal Residual Disease (MRD) Negativity Rate | Up to approximately 5 years
Number Of Participants With Adverse Events (AEs) | Up to approximately 5 years
Change From Baseline in the European Organization for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ-C30) | Up to approximately 5 years
  The EORTC QLQ-C30 is the most commonly used quality of life instrument in oncology trials. The QLQ-C30 consists of 30 questions incorporated into 5 functional domains physical, role, cognitive, emotional, and social), 9 symptom/other scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a single global Quality of Life (QoL)/global health status score. Items in the functional and symptom scale use raw participant response of 1 to 4, where 1 = "not at all" and 4 = "very much." The 2 global items contain responses ranging from 1 "very poor" to 7 "excellent." The recall period is 1 week. All domain scores are transformed in a range from 0 to 100, where a higher functional score indicates more favorable outcomes and a higher score on the symptom domains indicates a less favorable participant outcome. Stage 2 only.
Change From Baseline in the European Quality of Life Multiple Myeloma Module (EORTC QLQ-MY20) | Up to approximately 5 years
  The EORTC QLQ-MY20 is a 20-item myeloma module intended for use among participants varying in disease stage and treatment modality. Participants rate symptoms or problems on a scale from 1 to 4 where 1 = "not at all" and 4 = "very much." Stage 2 only.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (207):
- United States (34):
  - Local Institution - 0046, Mobile, Alabama
  - Local Institution - 0005, Cerritos, California
  - Local Institution - 0190, Irvine, California
  - Local Institution - 0187, Los Angeles, California
  - Local Institution - 0344, Santa Rosa, California
  - Local Institution - 0339, Stockton, California
  - Local Institution - 0279, Newark, Delaware
  - Local Institution - 0341, Fort Myers, Florida
  - Local Institution - 0342, St. Petersburg, Florida
  - Local Institution - 0340, West Palm Beach, Florida
  - Local Institution - 0348, Atlanta, Georgia
  - Local Institution - 0291, Atlanta, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Local Institution - 0289, Annapolis, Maryland
  - Local Institution - 0204, Boston, Massachusetts
  - Local Institution - 0346, Minneapolis, Minnesota
  - Local Institution - 0222, Little Silver, New Jersey
  - Local Institution - 0199, The Bronx, New York
  - Local Institution - 0322, Cleveland, Ohio
  - Local Institution - 0172, Columbus, Ohio
  - Local Institution - 0321, Providence, Rhode Island
  - Local Institution - 0338, Greer, South Carolina
  - Local Institution - 0349, Chattanooga, Tennessee
  - Local Institution - 0323, Nashville, Tennessee
  - Local Institution - 0337, Fort Worth, Texas
  - Local Institution - 0328, Houston, Texas
  - Local Institution - 0044, Houston, Texas
  - Local Institution - 0195, Temple, Texas
  - Local Institution - 0345, Norfolk, Virginia
  - Local Institution - 0343, Roanoke, Virginia
  - Local Institution - 0006, Tacoma, Washington
  - Local Institution - 0347, Vancouver, Washington
  - Local Institution - 0243, Morgantown, West Virginia
  - Local Institution - 0336, Marshfield, Wisconsin
- Argentina (6):
  - Local Institution - 0008, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0079, ABB, Buenos Aires F.D.
  - Local Institution - 0182, Rosario, Santa Fe Province
  - Local Institution - 0319, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0150, Buenos Aires
  - Local Institution - 0151, Córdoba
- Australia (10):
  - Local Institution - 0077, Camperdown, New South Wales
  - Local Institution - 0160, Gosford, New South Wales
  - Local Institution - 0263, Port Macquarie, New South Wales
  - Local Institution - 0078, St Leonards, New South Wales
  - Local Institution - 0026, Sydney, New South Wales
  - Local Institution - 0024, Adelaide, South Australia
  - Local Institution - 0131, Bendigo, Victoria
  - Local Institution - 0224, East Melbourne, Victoria
  - Local Institution - 0127, Heidelberg, Victoria
  - Local Institution - 0025, Melbourne, Victoria
- Austria (3):
  - Local Institution - 0266, Vienna, Vienna
  - Local Institution - 0020, Linz
  - Local Institution - 0017, Vienna
- Brazil (5):
  - Local Institution - 0121, Salvador, Estado de Bahia
  - Local Institution - 0076, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0085, São Paulo, São Paulo
  - Local Institution - 0075, Rio de Janeiro
  - Local Institution - 0073, São Paulo
- Bulgaria (3):
  - Local Institution - 0305, Plovdiv
  - Local Institution - 0309, Sofia
  - Local Institution - 0304, Sofia
- Canada (3):
  - Local Institution - 0183, Halifax, Nova Scotia
  - Local Institution - 0275, London, Ontario
  - Local Institution - 0184, Toronto, Ontario
- China (29):
  - Local Institution - 0318, Hefei, Anhui
  - Local Institution - 0061, Beijing, Beijing Municipality
  - Local Institution - 0057, Beijing, Beijing Municipality
  - Local Institution - 0056, Beijing, Beijing Municipality
  - Local Institution - 0123, Fuzhou, Fujian
  - Local Institution - 0138, Guangzhou, Guangdong
  - Local Institution - 0315, Guangzhou, Guangdong
  - Local Institution - 0051, Zhengzhou, Henan
  - Local Institution - 0066, Wuhan, Hubei
  - Local Institution - 0054, Wuhan, Hubei
  - Local Institution - 0071, Changsha, Hunan
  - Local Institution - 0103, Changsha, Hunan
  - Local Institution - 0180, Nanjing, Jiangsu
  - Local Institution - 0111, Nantong, Jiangsu
  - Local Institution - 0104, Suzhou, Jiangsu
  - Local Institution - 0069, Wuxi, Jiangsu
  - Local Institution - 0095, Nanchang, Jiangxi
  - Local Institution - 0052, Changchun, Jilin
  - Local Institution - 0096, Shenyang, Liaoning
  - Local Institution - 0176, Shenyang, Liaoning
  - Local Institution - 0060, Xi'an, Shaanxi
  - Local Institution - 0072, Jinan, Shandong
  - Local Institution - 0118, Shanghai, Shanghai Municipality
  - Local Institution - 0317, Shanghai, Shanghai Municipality
  - Local Institution - 0091, Tianjin, Tianjin Municipality
  - Local Institution - 0058, Kunming, Yunnan
  - Local Institution - 0050, Hangzhou, Zhejiang
  - Local Institution - 0115, Wenzhou, Zhejiang
  - Local Institution - 0059, Taiyuan
- Colombia (5):
  - Local Institution - 0153, Medellín, Antioquia
  - Local Institution - 0156, Valledupar, Cesar Department
  - Local Institution - 0154, Bogota, Cundinamarca
  - Local Institution - 0324, Piedecuesta, Santander Department
  - Local Institution - 0155, Cali
- Denmark (4):
  - Local Institution - 0032, Aarhus, Central Jutland
  - Local Institution - 0065, Roskilde, Region Sjælland
  - Local Institution - 0129, Odense, Region Syddanmark
  - Local Institution - 0125, Vejle
- Germany (14):
  - Local Institution - 0124, Ulm, Baden-Wurttemberg
  - Local Institution - 0330, Munich, Bavaria
  - Local Institution - 0333, Hanover, Lower Saxony
  - Local Institution - 0335, Dortmund, North Rhine-Westphalia
  - Local Institution - 0029, Kiel, Schleswig-Holstein
  - Local Institution - 0331, Jena, Thuringia
  - Local Institution - 0007, Berlin
  - Local Institution - 0102, Cologne
  - Local Institution - 0329, Dresden
  - Local Institution - 0334, Düsseldorf
  - Local Institution - 0015, Heidelberg
  - Local Institution - 0030, Leipzig
  - Local Institution - 0133, Nuremberg
  - Local Institution - 0014, Würzburg
- Greece (3):
  - Local Institution - 0136, Pátrai, Achaḯa
  - Local Institution - 0135, Athens, Attikí
  - Local Institution - 0134, Thessaloniki, Thessaloníki
- Local Institution - 0178, Hksar, Hong Kong
- Hungary (5):
  - Local Institution - 0036, Pécs, Baranya
  - Local Institution - 0043, Debrecen, Hajdú-Bihar
  - Local Institution - 0094, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Local Institution - 0042, Budapest
  - Local Institution - 0019, Budapest
- India (11):
  - Local Institution - 0167, Gurgaon, Haryana
  - Local Institution - 0161, Bengaluru, Karnataka
  - Local Institution - 0168, Mumbai, Maharashtra
  - Local Institution - 0171, Thane, Maharashtra
  - Local Institution - 0170, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0261, Mohali, Punjab
  - Local Institution - 0174, Chennai, Tamil Nadu
  - Local Institution - 0165, Hyderabad, Telangana
  - Local Institution - 0310, Hyderabad, Telangana
  - Local Institution - 0164, Hyderabad, Telangana
  - Local Institution - 0230, Chandigarh
- Israel (3):
  - Local Institution - 0264, Holon, Central District
  - Local Institution - 0267, Ẕerifin, Central District
  - Local Institution - 0277, Jerusalem
- Italy (8):
  - Local Institution - 0145, Meldola, Emilia-Romagna
  - Local Institution - 0143, Milan, Lombardy
  - Local Institution - 0142, Rozzano, Milano
  - Local Institution - 0189, Bologna
  - Local Institution - 0148, Catanzaro
  - Local Institution - 0147, Lecce
  - Local Institution - 0144, Pisa
  - Local Institution - 0146, Udine
- Japan (22):
  - Local Institution - 0269, Nagoya, Aichi-ken
  - Local Institution - 0214, Kashiwa, Chiba
  - Local Institution - 0210, Kitakyushu-shi, Fukuoka
  - Local Institution - 0211, Sapporo, Hokkaido
  - Local Institution - 0217, Higashiibaraki, Ibaraki
  - Local Institution - 0300, Kanazawa, Ishikawa-ken
  - Local Institution - 0209, Shiwa-gun Yahaba-cho, Iwate
  - Local Institution - 0234, Kamakura, Kanagawa
  - Local Institution - 0225, Koshigaya, Saitama
  - Local Institution - 0236, Itabashiku, Tokyo
  - Local Institution - 0219, Koto-ku, Tokyo
  - Local Institution - 0303, Chūō, Yamanashi
  - Local Institution - 0215, Chiba
  - Local Institution - 0226, Fukuoka
  - Local Institution - 0235, Fukuoka
  - Local Institution - 0220, Kumamoto
  - Local Institution - 0216, Kyoto
  - Local Institution - 0213, Nagasaki
  - Local Institution - 0212, Okayama
  - Local Institution - 0301, Osaka
  - Local Institution - 0241, Tokyo
  - Local Institution - 0218, Tokyo
- Netherlands (2):
  - Local Institution - 0113, Breda, North Brabant
  - Local Institution - 0194, Enschede
- Norway (3):
  - Local Institution - 0049, Bergen, Hordaland
  - Local Institution - 0112, Stavanger, Rogaland
  - Local Institution - 0081, Oslo
- Local Institution - 0316, San Juan, Puerto Rico
- Romania (5):
  - Local Institution - 0282, Bucharest, București
  - Local Institution - 0284, Brasov
  - Local Institution - 0302, Bucharest
  - Local Institution - 0287, Bucharest
  - Local Institution - 0306, Sibiu
- Singapore (2):
  - Local Institution - 0158, Singapore, Central Singapore
  - Local Institution - 0159, Singapore, Central Singapore
- South Korea (3):
  - Local Institution - 0238, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0239, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0240, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (10):
  - Local Institution - 0126, Badalona, Barcelona [Barcelona]
  - Local Institution - 0092, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0038, L'Hospitalet Del Llobregat, Barcelona [Barcelona]
  - Local Institution - 0200, Madrid, Madrid, Comunidad de
  - Local Institution - 0108, Majadahonda, Madrid, Comunidad de
  - Local Institution - 0201, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Local Institution - 0037, Valencia, Valenciana, Comunitat
  - Local Institution - 0107, Granada
  - Local Institution - 0047, Madrid
  - Local Institution - 0105, Málaga
- Taiwan (6):
  - Local Institution - 0274, Chiayi City, Chiayi
  - Local Institution - 0177, Kaohsiung Niao Sung Dist, Kaohsiung
  - Local Institution - 0012, Kaohsiung City
  - Local Institution - 0001, Taichung
  - Local Institution - 0002, Tainan
  - Local Institution - 0162, Taipei
- United Kingdom (6):
  - Local Institution - 0139, Plymouth, Devon
  - Local Institution - 0067, Cringleford, England
  - Local Institution - 0196, Glasgow, Glasgow City
  - Local Institution - 0273, Birmingham
  - Local Institution - 0080, Leeds
  - Local Institution - 0040, Taunton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05552976.html